CLINICAL TRIAL: NCT06828874
Title: A Prospective, Multicenter, Randomized, Blinded, Positive Parallel Control Study to Estimate the Efficacy and Safety of Levornidazole Disodium Phosphate for Injection in the Treatment of Postoperative Intra-Abdominal Infections Caused by Anaerobic Bacteria
Brief Title: A Study of Levornidazole Disodium Phosphate for Injection vs. Ornidazole in Treatment of Postoperative Intra-Abdominal Infections Caused by Anaerobic Bacteria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yangtze River Pharmaceutical Group Jiangsu Zilong Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Yangtze River Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YRPG-PMS-XR-RCT-2022-03
Record Dates: First submitted 2025-02-10; First posted 2025-02-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Intraabdominal Infections
MeSH Terms: conditions — Intraabdominal Infections | interventions — Injections; Ornidazole; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Drug: Levornidazole Disodium Phosphate for Injection
- Control Group (Active Comparator)
  Interventions: Drug: Ornidazole and Sodium Chloride Injection

INTERVENTIONS:
Drug: Levornidazole Disodium Phosphate for Injection — 1g，once daily, intravenously guttae for 4 to 7 days
  Arms: Experimental Group
Drug: Ornidazole and Sodium Chloride Injection — 0.5g at a time , 2 times per day, intravenously guttae for 4 to 7 days
  Arms: Control Group

SUMMARY:
Anaerobic infections are very common in clinical practice. Poor control of anaerobic infections in patients undergoing abdominal surgery may lead to the occurrence of complications. The aim of this study is to explore the efficacy and safety of Levornidazole Phosphate Disodium for Injection in the treatment of patients with postoperative intra-abdominal infections caused by anaerobic bacteria.

ELIGIBILITY:
Inclusion criteria：

Subjects who meet all of the following criteria may be enrolled in the study:

1. Age between 18 and 75 years old
2. Requires minimally invasive surgery (laparoscopic surgery or robotic-assisted surgery), open or percutaneous drainage surgery; Intra-abdominal infection caused by anaerobic bacteria as judged by the investigator, including purulent appendicitis, gangrene perforated appendicitis, periappendiceal abscess, gastric or duodenal perforation or rupture, jejunum, ileum, colorectal perforation or rupture, acute biliary tract infection and liver abscess; and meet at least one of the following two criteria: (1)At least two of the following four conditions must be met within 24 hours before surgery: abdominal pain, tenderness and fever (axillary temperature ≥ 37.5℃); white blood cell count ≥ 10×10^9/L; C-reactive protein above the upper limit of normal; procalcitonin (PCT)above the upper limit of normal;(2) Computed Tomography (CT) or ultrasound confirms the presence of intra-abdominal infection
3. Agree or plan to use the investigational drug for the first time within 24 hours postoperatively
4. The subjects voluntarily underwent the test and signed the informed consent form, and the process of signing the informed consent form was in line with Good Clinical Practice (GCP) guidelines

Exclusion criteria：

Subjects who meet any of the following criteria should be excluded from this study:

1. Those with known or suspected allergies to nitroimidazoles
2. Patients who have participated in other studies and used investigational drugs of other studies within 3 months prior to screening
3. Patients who are taking other medications or have other diseases that may interfere with the evaluation of the safety or effectiveness of the drug; Or patients who are at risk of serious drug interactions due to concomitant medications(such as warfarin, as well as medications with compatibility contraindications to levornidazole, including furbencillin sodium, nafcillin sodium, omeprazole, vorbizole, potassium sodium dehydroandrographolide succinate for injection, azlocillin sodium, etc.)
4. patients who have poor compliance and cannot complete the expected course of treatment and follow-up in the opinion of the investigator
5. Abnormal liver function (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times the upper limit of the normal value; for patients with acute biliary tract infection or combined liver abscess, it can be relaxed to > 3 times the upper limit of the normal value); or abnormal kidney function (creatinine clearance rate ≤ 60 mL/min/1.73 m² [Cockcroft - Gault formula])
6. Patients with serious primary diseases of important organs and systems such as cardiovascular, nervous system, endocrine system, hematopoietic system (such as heart failure, leukemia, uncontrolled diabetes, etc.), or those with malignant tumors
7. Women during pregnancy or lactation, or women of childbearing age with a positive pregnancy test result before the trial
8. Women of childbearing age and men who cannot take effective contraceptive measures during the trial period. The time limit is from the signing of the informed consent form to 3 months after the last dose
9. Patients with infections other than the abdomen (chronic infections that do not affect the evaluation of intra-abdominal infections [such as chronic rhinitis, chronic pharyngitis, etc.] can be included in this study)
10. Patients with multiple organ failure
11. Those who are considered by the investigator to be severely ill and need to be treated with other broad-spectrum antibiotics with anti-anaerobic effects (except for first/second/third generation cephalosporins, aztreonam, quinolones, aminoglycosides).
12. Those who have received antibiotic treatment within 48 hours before enrollment and randomization(except for single dose)
13. Those with positive test results for hepatitis B surface antigen, acquired immunodeficiency syndrome (AIDS) antibody, treponema pallidum antibody, and hepatitis C antibody
14. Patients with lesions of the brain and spinal cord, epilepsy, organ sclerosis, hematopoietic insufficiency, chronic alcoholism
15. Other patients who are not suitable to participate in this clinical study in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with clinical cure at Test of Cure (TOC) visit | 5 to 10 days post-therapy
  Clinical cure was defined as complete resolution of all symptoms and signs, including the return to normal of non - microbiological indicators such as preoperative imaging and laboratory tests. Symptoms and laboratory tests returned to normal using the following criteria: resolution or improvement of abdominal pain; Body temperature ≤ 37.5°C and white blood cell count < 10×10^9/L. persistent or incomplete resolution or worsening of symptoms and signs; or the development of new symptoms or signs and/or the use of other antimicrobial drugs against anaerobes was defined as clinically failure. The percentage of participants with clinical cure or clinical failure at TOC was summarized.

SECONDARY OUTCOMES:
Proportion of participants with clinical cure at End of Therapy (EOT) visit | Up to approximately Day 8
  Clinical cure was defined as complete resolution of all symptoms and signs, including the return to normal of non - microbiological indicators such as preoperative imaging and laboratory tests. Symptoms and laboratory tests returned to normal using the following criteria: resolution or improvement of abdominal pain; Body temperature ≤ 37.5°C and white blood cell count < 10×10^9/L.
Bacteriological efficacy at EOT visit | Up to approximately Day 8
  Bacteriological efficacy included eradication (absence of the baseline bacterial pathogen in a specimen appropriately obtained from the original site of infection) or presumed eradication (absence of material to culture in a participant who is assessed as a clinical cure). Bacteriological efficacy was evaluated only in cases where anaerobic cultures were positive for specimens obtained during baseline surgery. The percentage of participants with a favorable per-participant microbiological response of eradication or presumed eradication was reported for the EOT visit.
Comprehensive efficacy at EOT visit | Up to approximately Day 8
  Comprehensive efficacy was evaluated only in cases where anaerobic cultures were positive for specimens obtained during baseline surgery. It was an evaluation based on a combination of clinical and bacteriological results, and was divided into cured and ineffective. The former implied clinical cure with bacteria eradication or presumed eradication. The latter referred to clinical failure or bacterial non-eradication or presumed non-eradication, or both. The percentage of participants who were cured or ineffective was summarized for the EOT visit.
Bacteriological efficacy at TOC visit | 5 to 10 days post-therapy
  Bacteriological efficacy included eradication (absence of the baseline bacterial pathogen in a specimen appropriately obtained from the original site of infection) or presumed eradication (absence of material to culture in a participant who is assessed as a clinical cure). Bacteriological efficacy was evaluated only in cases where anaerobic cultures were positive for specimens obtained during baseline surgery. The percentage of participants with a favorable per-participant microbiological response of eradication or presumed eradication was reported for the TOC visit.
Comprehensive efficacy at TOC visit | 5 to 10 days post-therapy
  Comprehensive efficacy was evaluated only in cases where anaerobic cultures were positive for specimens obtained during baseline surgery. It was an evaluation based on a combination of clinical and bacteriological results, and was divided into cured and ineffective. The former implied clinical cure with bacteria eradication or presumed eradication. The latter referred to clinical failure or bacterial non-eradication or presumed non-eradication, or both. The percentage of participants who were cured or ineffective was summarized for the TOC visit.
Incidence of phlebitis during treatment | Up to approximately Day 7
  Phlebitis may be associated with intravenous infusion of highly irritating, high-concentration drugs, or prolonged use, and is one of the safety indicators. The percentage of participants who developed phlebitis was summarized during treatment.
Percentage of participants who experienced Adverse Events (AEs) | Up to Day 10 post-therapy
  An AE was any untoward medical occurrence in a participant administered a pharmaceutical product that did not necessarily have to have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. The percentage of participants who experienced AEs were summarized.

CONTACTS AND LOCATIONS:
Locations (32):
- China (32):
  - Chizhou People's Hospital, Chizhou, Anhui
  - Taihe County People's Hospital, Fuyang, Anhui
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Shaoyang University, Shaoyang, Hunan
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - Jiangyin People's Hospital, Wuxi, Jiangsu
  - Yixing People's Hospital, Wuxi, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Provincial Hospital of Traditional Chinese Medicine, Jinan, Shandong
  - Rizhao People's Hospital, Rizhao, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Dongyang People's Hospital, Jinhua, Zhejiang
  - Jinhua People's Hospital, Jinhua, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang